CLINICAL TRIAL: NCT05028192
Title: Mitochondria Preservation by Exercise Training: A Targeted Therapy for Cancer and Chemotherapy-induced Cachexia.
Acronym: MEx
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Turin, Italy (Other)
Collaborators: University of Padova (Other); Catholic University of the Sacred Heart (Other); University of Roma La Sapienza (Other)
Responsible Party: Sponsor
Other Study IDs: N. 98/2021
Record Dates: First submitted 2021-05-25; First posted 2021-08-31 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Cachexia; Rectal Cancer
MeSH Terms: conditions — Cachexia; Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Oblique or rectus abdominis muscle biopsy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Rectal cancer after neoadjuvant treatment: Rectal cancer patients, ycTNM stage II, III, and IV (AJCC 8th), clinically stratified in the pre-cachectic or cachectic stage according to Fearon K et al. definition. That will be subject to curative intent resection or palliative surgery through any approach (open, laparoscopic, or robotic).
  Interventions: Other: no intervention
- Control group: Patients who will undergo programmed abdominal surgery through any approach type for no neoplastic or inflammatory disease.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
This study aims to define the contribution of cancer and chemotherapy to muscle and systemic alterations that drive the onset of cachexia in rectal cancer patients and validate in human cancer cachexia (CC) the alterations in mitochondrial function and neuromuscular junction (NMJ) observed in the experimental models, thus providing the rationale for potential anti-cachexia strategies based on exercise and or exercise mimetics.

DETAILED DESCRIPTION:
This is a multicenter observational prospective cohort study in rectal cancer patients after neoadjuvant therapy (ycTNM) stage II, III, and IV (AJCC 8th edit), clinically stratified in the pre-cachectic or cachectic stage according to Fearon K et al. definition. That will be subject to curative or palliative surgery through any surgical approach. And a control subgroup of patients who will undergo any abdominal surgery type through any approach type for no neoplastic or inflammatory disease.

The study will take place in four Italian centers of colorectal surgery.

Will be run a preoperatory physical performance, and will be recorded the physical activity by wearing a SmartWatch.

The quantity of muscle will be estimated by the cross-sectional area (CSA) or the skeletal muscle area (SMA) from the magnetic resonance imaging (MRI) or computed tomography CT, respectively, and the Skeletal muscle index (SMI). The muscular quality will be studied by the mean skeletal muscle radiation attenuation (SMRA) and MRI proton density fat fraction (PDFF). All these parameters will be calculated by a radiologist from the preoperative MRI or CT imaging study.

The study includes the analysis of preoperatory inflammatory and nutritional biomarkers. And a muscular biopsy harvested by the surgeon from the rectum or oblique abdominal during rectal resection-palliative surgery. The sample will undergo morphological and structural studies using histology, immunohistochemical, immunofluorescence, biochemical, and molecular analyses.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed histopathological diagnosis of rectal adenocarcinoma ycTNM stage II, III, or IV (AJCC 8th).
* Patients treated with neoadjuvant therapy.
* Patients that will be subject to curative intent or palliative surgery through any approach (open, laparoscopic, or robotic).
* Ability to sign the informed consent.

Exclusion Criteria:

* Rectal cancer stage I or any stage without neoadjuvant therapy.
* Age < 18 and >75 years
* Long steroid treatment for any cause.
* Emergency setting.
* Co-existent inflammatory bowel disease.
* Inflammatory comorbidities (liver failure, diabetes, metabolic acidosis, acute and chronic renal failure, sepsis, AIDS, acute and chronic hepatitis, autoimmune disorders, and chronic obstructive pulmonary disease).
* Healthy volunteers.
* Other (simultaneous) neoplastic disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from all participating centers older than 18 years, males or females, with the primary diagnosis of rectal cancer ycTNM stage II, III or IV (American Joint Committee on Cancer 8th edition), who undergone neoadjuvant therapy. Clinically stratified in the pre-cachectic or cachectic stage according to Fearon K et al. definition. That will be subject to low or ultralow anterior resection, abdominoperineal resection or palliative surgery through any approach (open, laparoscopic or robotic).
Sampling Method: Probability Sample
Enrollment: 144 (Estimated)
Dates: Start 2021-09-27 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Physical function | Preoperative.
  Determinate by the short physical performance battery (SPPB) Score, a series of tests used to evaluate lower extremity function and mobility in older people. Scores are assigned according to performance, with an overall maximum score of 12. A cut off score < 10 indicates mobility disability and cut point: ≤ 8 points for diagnosing of severe sarcopenia
Physical activity-Subjective Measurement | Preoperative
  Determinate by the physical activity scale for the elderly (PASE) Score, the overall score ranging from 0 to 793, higher scores indicated greater physical activity
Physical activity-Objective Measurement (step count) | Preoperative.
  Determinate by the average daily step count (total number of steps/14 days) recorded by wearing a Smart Watch for two weeks on consecutive days.
Physical activity-Objective Measurement (sleep) | Preoperative.
  Determinate by the average of daily sleep duration(total minutes of sleep/ 14 days) recorded by wearing a Smart Watch for two weeks on consecutive days.
Physical activity-Objective Measurement (sedentary time) | Preoperative.
  Determinate by the average daily sedentary time (total minutes of inactivity/14 days) recorded by wearing a Smart Watch for two weeks on consecutive days.
Physical activity-Objective Measurement (active time) | Preoperative.
  Determinate by the average daily active time (total duration of activity in minutes/14 days) recorded by wearing a Smart Watch for two weeks on consecutive days.
Muscular quantity | Preoperative.
  Determinate by the Skeletal muscle index (SMI) = skeletal muscle area or cross-sectional area at L4-L5 (cm2)/height2(m2) from the preoperative magnetic resonance imaging.
Muscular quality (muscle fat content) by magnetic resonance imaging | Preoperative.
  Determinate by the proton density fat fraction (PDFF) of paraspinal muscles at L4-L5
Nutritional status - Albumin | Preoperative.
  Blood levels of albumin (g/dL).
Nutritional status - Prealbumin | Preoperative.
  Blood levels of prealbumin(mg/dL).
Nutritional status - transferrin | Preoperative.
  Blood levels of transferrin(mg/dL).
General health marker- hemoglobin | Preoperative.
  Blood levels of Hemoglobin (g/L).
Inflammatory status-White blood cells count | Preoperative.
  White blood cells count (10^/L).
Inflammatory status - C-reactive protein | Preoperative.
  Blood levels of C-reactive protein (mg/dL).
Muscle wasting- creatine kinase | Preoperative.
  Blood levels of creatine kinase (U/L).
Morphometric analysis of skeletal muscle | within 30 postoperative days.
  Description of the dimension and type of muscular fibers from an abdominal wall muscle biopsy harvested intraoperatively.
Molecular analysis of skeletal muscle | within 60 postoperative days.
  Characterization of molecular signatures associated with Neo-adjuvant Chemotherapy and rectal cancer by comparing molecular profiles of a muscular biopsies harvested intraoperatively.
Muscle protein metabolism | within 60 postoperative days.
  Muscle-specific ubiquitin-ligases expression, mitophagy cargo shuttle, fusion-fission machinery, and mitochondrial biogenesis will be assayed from a muscular biopsy harvested intraoperatively.

SECONDARY OUTCOMES:
Overall survival | 3 years after surgery.
  to describe the percentage of participants who are alive three years after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Degiuli, Prof., Study Chair — Università degli studi di Torino- Surgical Oncology and Digestive Surgery
Locations (1):
- Ospedale San Luigi Gonzaga, Orbassano, Turin, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dev R. Measuring cachexia-diagnostic criteria. Ann Palliat Med. 2019 Jan;8(1):24-32. doi: 10.21037/apm.2018.08.07. Epub 2018 Sep 7. PMID 30525765
- [Background] Fearon K, Strasser F, Anker SD, Bosaeus I, Bruera E, Fainsinger RL, Jatoi A, Loprinzi C, MacDonald N, Mantovani G, Davis M, Muscaritoli M, Ottery F, Radbruch L, Ravasco P, Walsh D, Wilcock A, Kaasa S, Baracos VE. Definition and classification of cancer cachexia: an international consensus. Lancet Oncol. 2011 May;12(5):489-95. doi: 10.1016/S1470-2045(10)70218-7. Epub 2011 Feb 4. PMID 21296615
- [Background] Freire PP, Fernandez GJ, Cury SS, de Moraes D, Oliveira JS, de Oliveira G, Dal-Pai-Silva M, Dos Reis PP, Carvalho RF. The Pathway to Cancer Cachexia: MicroRNA-Regulated Networks in Muscle Wasting Based on Integrative Meta-Analysis. Int J Mol Sci. 2019 Apr 22;20(8):1962. doi: 10.3390/ijms20081962. PMID 31013615
- [Background] Baracos VE. Skeletal muscle anabolism in patients with advanced cancer. Lancet Oncol. 2015 Jan;16(1):13-4. doi: 10.1016/S1470-2045(14)71185-4. Epub 2014 Dec 16. No abstract available. PMID 25524803
- [Background] Wiegert EVM, de Oliveira LC, Calixto-Lima L, Borges NA, Rodrigues J, da Mota E Silva Lopes MS, Peres WAF. Association between low muscle mass and survival in incurable cancer patients: A systematic review. Nutrition. 2020 Apr;72:110695. doi: 10.1016/j.nut.2019.110695. Epub 2019 Dec 7. PMID 32007806
- [Background] Cruz-Jentoft AJ, Bahat G, Bauer J, Boirie Y, Bruyere O, Cederholm T, Cooper C, Landi F, Rolland Y, Sayer AA, Schneider SM, Sieber CC, Topinkova E, Vandewoude M, Visser M, Zamboni M; Writing Group for the European Working Group on Sarcopenia in Older People 2 (EWGSOP2), and the Extended Group for EWGSOP2. Sarcopenia: revised European consensus on definition and diagnosis. Age Ageing. 2019 Jul 1;48(4):601. doi: 10.1093/ageing/afz046. No abstract available. PMID 31081853
- [Background] Penet MF, Bhujwalla ZM. Cancer cachexia, recent advances, and future directions. Cancer J. 2015 Mar-Apr;21(2):117-22. doi: 10.1097/PPO.0000000000000100. PMID 25815852
- [Background] Codari M, Zanardo M, di Sabato ME, Nocerino E, Messina C, Sconfienza LM, Sardanelli F. MRI-Derived Biomarkers Related to Sarcopenia: A Systematic Review. J Magn Reson Imaging. 2020 Apr;51(4):1117-1127. doi: 10.1002/jmri.26931. Epub 2019 Sep 13. PMID 31515891